CLINICAL TRIAL: NCT04323527
Title: Efficacy and Safety of Chloroquine Diphosphate for the Treatment of Hospitalized Patients With Severe Acute Respiratory Syndrome Secondary to SARS-CoV2: a Phase IIb, Double-blind, Randomized Adaptive Clinical Trial
Brief Title: Chloroquine Diphosphate for the Treatment of Severe Acute Respiratory Syndrome Secondary to SARS-CoV2
Acronym: CloroCOVID19
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fundação de Medicina Tropical Dr. Heitor Vieira Dourado (Other)
Collaborators: Marcus Vinícius Guimarães de Lacerda (Unknown); Mayla Gabriela Silva Borba (Unknown); Wuelton Marcelo Monteiro (Unknown); Gisely Cardoso de Melo (Unknown); Fernando Fonseca de Almeida e Val (Unknown); Felipe Gomes Naveca (Unknown); Maria Paula Gomes Mourão (Unknown); Ludmila Abrahão Hajjar (Unknown); Jorge Souza Mendonça (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAAE: 30152620.1.0000.0005
Record Dates: First submitted 2020-03-19; First posted 2020-03-26 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: SARS-CoV Infection; Severe Acute Respiratory Syndrome (SARS) Pneumonia
Keywords: COVID-19; SARS-CoV Infection; Severe Acute Respiratory Syndrome (SARS) Pneumonia; Chloroquine Diphosphate; Clinical trial
MeSH Terms: conditions — Severe Acute Respiratory Syndrome; Pneumonia; COVID-19 | interventions — chloroquine diphosphate; Chloroquine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Low Dose Chloroquine Diphosphate (5 days) (Study stage 1) - Clorocovid 1 (Active Comparator): Low dose chloroquine group consists of 450 mg bid (3 tablets of 150 mg + 1 placebo tablet, every 12 hours) on D1, 3x150mg tablets + 1 placebo followed by 4 placebo tablets 12h later from D2 to D5, and 4 placebo tablets every 12 hours, D6-D10 . Oral administration or via nasogastric tube in case of orotracheal intubation. (this was the first stage of the original study and was approved by the Brazilian IRB on 23/March/2020).
  Interventions: Drug: Chloroquine diphosphate
- High Dose Chloroquine Diphosphate (10 days) (Study stage 1) - Clorocovid 1 (Active Comparator): High dose chloroquine group consists of 600 mg bid (4 tablets of 150 mg, every 12 hours) for 10 days. Oral administration or via nasogastric tube in case of orotracheal intubation. (this was the first stage of the original study and was approved by the Brazilian IRB on 23/March/2020).
  Interventions: Drug: Chloroquine diphosphate
- Placebo (5 days) (Study stage 2) - Clorocovid 3 (Placebo Comparator): Placebo group consists of 3 placebo tablets bid (day 1), and 3 placebo tablets once daily from D2 to D5. Oral administration or via a nasogastric tube in case of orotracheal intubation. (this was a second stage of the original study and was approved by the Brazilian IRB on 03/May/2020).
  Interventions: Drug: Chloroquine diphosphate
- Low Dose Chloroquine Diphosphate (5 days) (Study stage 2) - Clorocovid 3 (Active Comparator): Low dose chloroquine group consisted of 450 mg bid (3 tablets of 150 mg) on D1, and 3x150mg tablet once daily from D2 to D5. Oral administration or via a nasogastric tube in case of orotracheal intubation. (this was a second stage of the original study and was approved by the Brazilian IRB on 03/May/2020).
  Interventions: Drug: Chloroquine diphosphate

INTERVENTIONS:
Drug: Chloroquine diphosphate — 150mg chloroquine diphosphate tablets. Note: Tablets used in the study were Chloroquine Diphosphate (produced by Farmanguinhos/Fiocruz), and the dosing stated in the clinicaltrials.gov refers to chloroquine base (in mg).
  Other Names: chloroquine

SUMMARY:
In December 2019, the Municipal Health Committee of Wuhan, China, identified an outbreak of viral pneumonia of unknown cause. This new coronavirus was called SARS-CoV-2 and the disease caused by that virus, COVID-19. Recent numbers show that 222,643 infections have been diagnosed with 9115 deaths, worldwide. Currently, there are no approved therapeutic agents available for coronaviruses. In this scenario, the situation of a global public health emergency and evidence about the potential positive effect of chloroquine (CQ) in most coronaviruses, including SARS-CoV-1, and recent data on small trials on SARS-CoV-2, the investigators intend to investigate the efficacy and the safety of CQ diphosphate in the treatment of hospitalized patients with severe acute respiratory syndrome in the scenario of SARS-CoV2. Preliminary in vitro studies and uncontrolled trials with low number of patients of CQ repositioning in the treatment of COVID-19 have been encouraging. The main hypothesis is that CQ diphosphate will reduce mortality in 50% in those with severe acute respiratory syndrome infected by the SARS-COV2. Therefore, the main objective is to assess whether the use of chloroquine diphosphate reduces mortality by 50% in the study population. The primary outcome is mortality in day 28 of follow-up. According to local contingency plan, developed by local government for COVID-19 in the State of Amazonas, the Hospital Pronto-Socorro Delphina Aziz, located in Manaus, is the reference unit for the admission of serious cases of the new virus. The unit currently has 50 ICU beds, with the possibility of expanding to 335 beds, if needed. The hospital also has trained multiprofessional human resources and adequate infrastructure. In total, 440 participants (220 per arm) will receive either high dose chloroquine 600 mg bid regime (4x150 mg tablets, every 12 hours, D1-D10) or low dose chloroquine 450mg bid regime (3x150mg tablets + 1 placebo tablet every 12 hours on D1, 3x150mg tablets + 1 placebo followed by 4 placebo tablets 12h later from D2 to D5, and 4 placebo tablets every 12 hours, D6-D10). Placebo tablets were used to standardize treatment duration and blind research team and patients. All drugs administered orally (or via nasogastric tube in case of orotracheal intubation). Both intervention and placebo drugs will be produced by Farmanguinhos. Clinical and laboratory data during hospitalization will be used to assess efficacy and safety outcomes.

ELIGIBILITY:
Inclusion criteria:

1. Male and female participants aged over 18 years old
2. Hospitalized
3. presenting:

   * respiratory rate higher than 24 breathing incursions per minute AND/OR
   * heart rate higher than 125 beats per minute (in the absence of fever) AND/OR
   * peripheral oxygen saturation lower than 90% in ambient air AND/OR
   * shock (defined as mean arterial pressure less than 65 mmHg, requiring vasopressor or oliguria or lowering level of consciousness)

Exclusion Criteria:

• None.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 278 (Actual)
Dates: Start 2020-03-23 (Actual); Primary Completion 2020-05-07 (Actual); Study Completion 2020-06-07 (Actual)

PRIMARY OUTCOMES:
Mortality rate reduction of 50% by day 28 | 28 days after randomization
  proportion of deaths at day 28 between groups compared

SECONDARY OUTCOMES:
Absolute mortality on days 7 and 14 | 7 and 14 days after first dose
  number of deaths at days 7 and 14 between groups compared
Improvement in overall subject's clinical status assessed in standardized clinical questionnaires on days 14 and 28 | 14 and 28 days after first dose
  clinical status
Improvement in daily clinical status assessed in standardized clinical questionnaires during hospitalization | during and after intervention, up to 28 days
  clinical status
Duration of supplemental oxygen (if applicable) | during and after intervention, up to 28 days
  supplemental oxygen
Duration of mechanical ventilation (if applicable) | during and after intervention, up to 28 days
  mechanical ventilation
Absolute duration of hospital stay in days | during and after intervention, up to 28 days
  hospitalization
Prevalence of grade 3 and 4 adverse events | during and after intervention, up to 28 days
  adverse events grade 3 and 4
Prevalence of serious adverse events | during and after intervention, up to 28 days
  adverse events
Change in serum creatinine level | during and after intervention, up to 28 days
  increase or decrease in serum creatinine compared to baseline
Change in serum troponin I level | during and after intervention, up to 28 days
  increase or decrease in serum troponin I compared to baseline
Change in serum aspartate aminotransferase level | during and after intervention, up to 28 days
  increase or decrease in serum aspartate aminotransferase compared to baseline
Change in serum CK-MB level | during and after intervention, up to 28 days
  increase or decrease in serum aspartate aminotransferase compared to baseline
Change in detectable viral load in respiratory tract swabs | during and after intervention, up to 28 days
  virus clearance from respiratory tract secretion
Viral concentration in blood samples | during and after intervention, up to 28 days
  viremia in blood detected through RT-PCR
Absolute number of causes leading to participant death (if applicable) | during and after intervention, up to 28 days
  death

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital e Pronto Socorro Delphina Rinaldi Abdel Aziz, Manaus, Amazonas, Brazil

IPD SHARING:
Plan to Share IPD: Yes
all patient data will be shared after study publication
Supporting Information: Study Protocol, SAP, CSR
Time Frame: after study publication
Access Criteria: upon request to researchers

REFERENCES:
- [Derived] Erratum: Correlation between clinical and pathological findings of liver injury in 27 patients with lethal COVID-19 infections in Brazil. Hepatol Commun. 2024 Jun 27;8(7):e0492. doi: 10.1097/HC9.0000000000000492. eCollection 2024 Jul 1. No abstract available. PMID 38934714
- [Derived] Borba MGS, Val FFA, Sampaio VS, Alexandre MAA, Melo GC, Brito M, Mourao MPG, Brito-Sousa JD, Baia-da-Silva D, Guerra MVF, Hajjar LA, Pinto RC, Balieiro AAS, Pacheco AGF, Santos JDO Jr, Naveca FG, Xavier MS, Siqueira AM, Schwarzbold A, Croda J, Nogueira ML, Romero GAS, Bassat Q, Fontes CJ, Albuquerque BC, Daniel-Ribeiro CT, Monteiro WM, Lacerda MVG; CloroCovid-19 Team. Effect of High vs Low Doses of Chloroquine Diphosphate as Adjunctive Therapy for Patients Hospitalized With Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) Infection: A Randomized Clinical Trial. JAMA Netw Open. 2020 Apr 24;3(4):e208857. doi: 10.1001/jamanetworkopen.2020.8857. PMID 32330277